CLINICAL TRIAL: NCT06901752
Title: Effectiveness of Kinesiotaping in Adolescent Idiopathic Scoliosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, MD, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAEK-11/12.02.2025.51
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Scoliosis Idiopathic Adolescent
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Research Group (Active Comparator): In addition to the regular exercise program, kinesio taping will be applied to patients diagnosed with Adolescent Idiopathic Scoliosis. Kinesio taping will be applied for 5 days on and 2 days off for 4 weeks.
  Interventions: Procedure: Kinesiotaping; Behavioral: Exercise
- Control Group (Placebo Comparator): Patients diagnosed with Adolescent Idiopathic Scoliosis will continue their regular exercise program. No intervention will be applied.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Procedure: Kinesiotaping — Kinesio Taping Method is a therapeutic tool utilised by rehabilitation specialists in all programs (paediatric, geriatric, orthopaedic, neurological, oncology and others) and levels of care (acute care,inpatient rehabilitation,outpatient, home care and Day Rehab). The idea of using elastic tape to mimic the therapist's hands was first presented by Dr Kenzo Kase in the 1970s. Since then, it became the modality used in pain management, soft tissue injury, tissues and joints malalignment, oedema, and more. Kinesio Taping Method utilises four types of Kinesio Tex Tapes, each with specific properties designed for use on fragile, sensitive skin or applied with higher tensions. Kinesio Taping Method has also effectively treated animals and two special tapes are used: Kinesio Equine and Kinesio Canine. Kinesio Tex Tape contains either 100% cotton and elastic fibres or a blend of polyester and cotton with elastic fibres. The latter is preferable for Kinesio Taping application on sensitive skin
  Arms: Research Group
Behavioral: Exercise — Cat Camel Exercise, Bridge Exercise, Lateral Flexion, Cross Walking, Ipsilateral and Contralateral Stretching Exercises

SUMMARY:
The effectiveness of kinesiotaping application in addition to exercise in Adolescent Idiopathic Scoliosis will be compared on the pain level with the numerical rating scale, the Cobb angle and scoliometer measurements, the quality of life with the Scoliosis Research Association-22 quality of life scale, and the patient's visual perception level with the Walter Reed visual assessment scale. Research Group: In addition to the regular exercise program, kinesio taping will be applied to patients diagnosed with Adolescent Idiopathic Scoliosis. Kinesio taping will be applied for 5 days on and 2 days off for 4 weeks. Control Group: Patients diagnosed with Adolescent Idiopathic Scoliosis will continue their regular exercise program. No intervention will be applied. Patients will be evaluated before and 3 months after treatment in terms of pain level with numerical rating scale, Cobb angle measurement and Scoliometer measurement, quality of life with Scoliosis Research Association-22 quality of life scale and Walter Reed visual assessment scale.

ELIGIBILITY:
Inclusion Criteria:

* Being under follow-up with the diagnosis of Adolescent Idiopathic Scoliosis
* Having a Cobb angle between 10-25 degrees
* Being willing to participate in the study
* Having thoracic C scoliosis

Exclusion Criteria:

* Having a spinal curvature of more than 25 degrees
* Presence of cardiopulmonary disease and musculoskeletal deformity that will prevent exercise
* Having an open wound in the area where kinesio taping will be applied or being allergic to the tape application
* Presence of S scoliosis

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Cobb Angle Measurement | 3 months
Scoliometer Measurement | 3 months

SECONDARY OUTCOMES:
Scoliosis Research Society-22 Test | 3 months
walter reed visual assessment scale | 3 months